CLINICAL TRIAL: NCT02431351
Title: A Phase 2, Open-Label, Single Arm Study Evaluating the Efficacy and Safety of the Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Erythropoietin (EPO)-Refractory Lower-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Efficacy & Safety Study of KPT-330 in Erythropoietin-Refractory Lower-Risk Myelodysplastic Syndrome Patients
Acronym: SIER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial never opened.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-014
Record Dates: First submitted 2015-04-27; First posted 2015-05-01 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: KPT-330; Karyopharm; Selinexor; SIER; Myelodysplastic Syndrome (MDS); Erythropoietin (EPO); Refractory
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selinexor (Experimental): 60 mg once weekly
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — 60 mg on Day 1 of each week for a 4 week cycle, given for ≥6 cycles.
  Other Names: KPT-330

SUMMARY:
This is an open-label study designed to evaluate the safety and efficacy of the selective inhibitor of nuclear export (SINE) compound, Selinexor given orally to patients with transfusion-dependent, EPO-refractory lower-risk MDS (Low risk and Intermediate-1 as defined by IPSS).

DETAILED DESCRIPTION:
This is a single-arm, open-label, study designed to evaluate the safety and efficacy of the selective inhibitor of nuclear export (SINE) compound, Selinexor given orally to patients with transfusion-dependent, EPO-refractory lower-risk MDS (Low risk and Intermediate-1 as defined by IPSS). Patients will be dosed at the clinic on clinic visit days and received Selinexor for dosing at home on additional days.

Patients will be evaluated for disease response according to the 2006 IWG response criteria for MDS. This includes evaluation for altering the natural history of disease, cytogenic response hematologic improvement, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Low risk or Intermediate-1 risk MDS with any cytogenetic abnormalities (according to the IPSS criteria); patients must have bone marrow biopsy/aspiration or tumor tissue available from within 1 month prior to first dose or collected during the Screening period.
* Patients >18 years at Screening who are not candidates for hematopoietic cell transplantation.
* Received 1 prior line of treatment; typically erythroid-stimulating agents (ESAs).
* Red blood cell (RBC) transfusion-dependent anemia while treated with or after discontinuation of EPO. Transfusion dependence is defined as the requirement for at least 2 units of RBCs transfused during the 8 weeks prior to study initiation.

Exclusion Criteria:

* Use of recombinant EPO within 8 weeks prior to screening.
* Patient has a concurrent active malignancy or prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma of the skin and in situ of the cervix) unless free of disease for at least 1 year.
* Unstable cardiovascular function:

  * Symptomatic ischemia,
  * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic Left anterior fascicular block/Right bundle branch block (LAFB/RBBB) will not be excluded), or
  * Congestive heart failure (CHF) New York Heart Association (NYHA) Class ≥3, or myocardial infarction (MI) within 3 months.
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
* Active bleeding Grade 3-4, in the last 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Hematologic improvement (based on the 2006 International Working Group (IWG) response criteria) | 6 months
  Hematologic improvement in erythroid, platelet, and neutrophil counts, evaluated based on the 2006 International Working Group (IWG) response criteria for MDS.

SECONDARY OUTCOMES:
Overall response rate | 6 months
  Overall response is defined as complete remission (CR) or partial remission (PR).
Quality of Life (QOL-E) MDS Questionnaire) | 6 months
  Evaluate quality of life using the Quality of Life-E (QOL-E) MDS Questionnaire